CLINICAL TRIAL: NCT05839067
Title: Supporting Physical & Mental Health in Rural Veterans With Heart Failure (CARE-HF)
Brief Title: Supporting Health in Veterans With Heart Failure
Acronym: CARE-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lucinda Graven, Associate Professor, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00003764
Record Dates: First submitted 2023-04-10; First posted 2023-05-03 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
Keywords: heart failure; problem-solving; Veterans; self-care; quality of life; depression; anxiety; stress; symptoms; resilience
MeSH Terms: conditions — Heart Failure; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 100 participants will be trained to use a 5-step theoretically driven problem-solving process to manage heart failure problems experienced in the home.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CARE-HF (Experimental): The problem-solving intervention will be led by a registered nurse. Participants will receive a program manual containing examples of common HF-related problems experienced by heart failure patients and suggested management strategies, with some strategies tailored to the rural sociocultural context. The nurse will lead participants in a card sorting task intended to help participants prioritize current HF-related problems and will guide participants in developing management strategies for the highest priority problem(s). Participants will utilize these strategies until the next session at which time the nurse will guide participants in evaluating the effectiveness of chosen strategies. The iterative process then begins again. Participants will receive 7 follow-up telephone sessions with the nurse. In the intervention, the nurse will focus on problems related to self-care, disease management, mental health, and quality of life, including those specific to the rural population.
  Interventions: Behavioral: Care-HF

INTERVENTIONS:
Behavioral: Care-HF — Participants will be trained to use a 5-step problem-solving process based on the Theory of Social Problem-Solving (TSPS) to manage HF-related problems over 12-weeks. The core belief of TSPS is effective problem-solving requires a positive problem orientation (i.e., viewing problems as a challenge versus a threat) and elicits rational problem-solving versus avoidance or impulsivity/carelessness. Problem-solving follows from a positive problem orientation and involves accurate problem identification, generation of appropriate potential solutions, active decision-making, and solution implementation and evaluation. The goal of this intervention is to move participants toward a positive problem orientation and use of rational problem-solving strategies that support greater physical and mental health.

SUMMARY:
This study will test the effectiveness of a culturally-sensitive, telephone-based, tailored problem-solving intervention to improve physical and mental health in Veterans with heart failure (HF). Veterans will be recruited from VA clinics throughout the United States. As a component of this study, Veterans will partner with a registered nurse for a 12-week telehealth program that includes 8 telephone sessions. Follow-up data will be collected at 3-months (post intervention) and 6-, 12-, and 18-months to examine sustainability of intervention effect.

DETAILED DESCRIPTION:
The long-term goal of this research is to support physical and mental health of Veterans with heart failure and enrich rehabilitation and independent living by enhancing disease self-management and coping processes in the home.

Study objectives include: (1) Evaluate the feasibility of recruitment and enrollment processes, attrition, and program acceptability in a sample of Veterans with HF; (2) Evaluate program effectiveness on study outcomes (i.e., self-care, symptoms, depression, anxiety, quality of life, stress, resilience, coping, and healthcare utilization); and (3) examine the sustainability of intervention effect.

This study will be guided by quantitative inquiry and include a single-group, repeated measures design. A sample size of 100 participants is desired based on a power analysis for repeated measures ANOVA with 5 time points, alpha level of .05, a medium effect size (f = 0.25), and 80% power, plus oversampling for potential attrition (20%). Following verbal informed consent via telephone, all participants will complete baseline data collection which will include a Sociodemographic and Clinical Survey, the Interpersonal Support Evaluation List - 12 (ISEL), the Social Problem-Solving Inventory Revised-Short (SPSIRs), the Self-care of Heart Failure Index (SCHFI, v 7.2), the Heart Failure Symptom Survey (HFSS), the Patient Health Questionnaire-9 (PHQ-9), the Generalized Anxiety Disorder (GAD) scale, the Minnesota Living with Heart Failure Questionnaire (MLHFQ), the Perceived Stress Scale (PSS), the 5x5 Resilience Scale, the Brief COPE, and a healthcare utilization survey.

All participants will participate in a tailored problem-solving intervention designed to help manage heart failure-related problems experienced in the home over 12 weeks (Weeks 1-4, 6, 8, 10, 12). Follow-up data collection will occur at 3-months (post-intervention) and 6-, 12-, and 18-months. Quantitative data on study variables will be collected using the following self-report surveys: SPSIRs, SCHFI, HFSS, PHQ-9, GAD, MLHFQ, PSS, 5x5 Resilience scale, Brief COPE, and healthcare utilization. All data will be collected by a trained research assistant who will collect study data over the telephone and mark participants answers on a computerized data spreadsheet. Possible treatment effectiveness on heart failure self-care, heart failure symptoms, healthcare utilization, depression, anxiety, quality of life, stress, resilience, coping, and differences among subgroups over the study period will be examined using multilevel modeling.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* US Veteran
* Diagnosed with heart failure (reduced or preserved ejection fraction)
* Able to read, speak, and understand English
* Reliable telephone access

Exclusion Criteria:

• History of cognitive dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Heart Failure Self-care | baseline
  Self-care maintenance, management, and confidence will be self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 7.0. Items pertain to treatment adherence and self-monitoring. Scores are standardized (0-100), with higher scores suggesting better self-care maintenance. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Heart Failure Self-care | 3-months
  Self-care maintenance, management, and confidence will be self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 7.0. Items pertain to treatment adherence and self-monitoring. Scores are standardized (0-100), with higher scores suggesting better self-care maintenance. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Heart Failure Self-care | 6-months
  Self-care maintenance, management, and confidence will be self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 7.0. Items pertain to treatment adherence and self-monitoring. Scores are standardized (0-100), with higher scores suggesting better self-care maintenance. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Heart Failure Self-care | 12-months
  Self-care maintenance, management, and confidence will be self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 7.0. Items pertain to treatment adherence and self-monitoring. Scores are standardized (0-100), with higher scores suggesting better self-care maintenance. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Heart Failure Self-care | 18-months
  Self-care maintenance, management, and confidence will be self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 7.0. Items pertain to treatment adherence and self-monitoring. Scores are standardized (0-100), with higher scores suggesting better self-care maintenance. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Heart Failure Symptoms | baseline
  Symptoms of HF will be assessed using the Heart Failure Symptom Survey (HFSS). This survey contains 14 symptoms commonly experienced by those with HF. Participants rate each symptom according to 4 domains (i.e., frequency, severity, interference with physical activity, and interference with enjoyment of life) based upon the last 7 days. Higher scores indicate more of the respective domain in relation to the particular symptom.
Heart Failure Symptoms | 3-months
  Symptoms of HF will be assessed using the Heart Failure Symptom Survey (HFSS). This survey contains 14 symptoms commonly experienced by those with HF. Participants rate each symptom according to 4 domains (i.e., frequency, severity, interference with physical activity, and interference with enjoyment of life) based upon the last 7 days. Higher scores indicate more of the respective domain in relation to the particular symptom.
Heart Failure Symptoms | 6-months
  Symptoms of HF will be assessed using the Heart Failure Symptom Survey (HFSS). This survey contains 14 symptoms commonly experienced by those with HF. Participants rate each symptom according to 4 domains (i.e., frequency, severity, interference with physical activity, and interference with enjoyment of life) based upon the last 7 days. Higher scores indicate more of the respective domain in relation to the particular symptom.
Heart Failure Symptoms | 12-months
  Symptoms of HF will be assessed using the Heart Failure Symptom Survey (HFSS). This survey contains 14 symptoms commonly experienced by those with HF. Participants rate each symptom according to 4 domains (i.e., frequency, severity, interference with physical activity, and interference with enjoyment of life) based upon the last 7 days. Higher scores indicate more of the respective domain in relation to the particular symptom.
Heart Failure Symptoms | 18-months
  Symptoms of HF will be assessed using the Heart Failure Symptom Survey (HFSS). This survey contains 14 symptoms commonly experienced by those with HF. Participants rate each symptom according to 4 domains (i.e., frequency, severity, interference with physical activity, and interference with enjoyment of life) based upon the last 7 days. Higher scores indicate more of the respective domain in relation to the particular symptom.
Depression | baseline
  Depression will be measured using the Patient Health Questionnaire-9 (PHQ-9). A PHQ-9 score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression.
Depression | 3-months
  Depression will be measured using the Patient Health Questionnaire-9 (PHQ-9). A PHQ-9 score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression.
Depression | 6-months
  Depression will be measured using the Patient Health Questionnaire-9 (PHQ-9). A PHQ-9 score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression.
Depression | 12 months
  Depression will be measured using the Patient Health Questionnaire-9 (PHQ-9). A PHQ-9 score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression.
Depression | 18 months
  Depression will be measured using the Patient Health Questionnaire-9 (PHQ-9). A PHQ-9 score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression.
Anxiety | baseline
  Anxiety will be measured using the Generalized Anxiety Disorder (GAD) scale. Scores are totaled and indicate the level of anxiety. Score 0-4: Minimal Anxiety. Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety.
Anxiety | 3-months
  Anxiety will be measured using the Generalized Anxiety Disorder (GAD) scale. Scores are totaled and indicate the level of anxiety. Score 0-4: Minimal Anxiety. Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety.
Anxiety | 6-months
  Anxiety will be measured using the Generalized Anxiety Disorder (GAD) scale. Scores are totaled and indicate the level of anxiety. Score 0-4: Minimal Anxiety. Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety.
Anxiety | 12-months
  Anxiety will be measured using the Generalized Anxiety Disorder (GAD) scale. Scores are totaled and indicate the level of anxiety. Score 0-4: Minimal Anxiety. Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety.
Anxiety | 18-months
  Anxiety will be measured using the Generalized Anxiety Disorder (GAD) scale. Scores are totaled and indicate the level of anxiety. Score 0-4: Minimal Anxiety. Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety.

SECONDARY OUTCOMES:
Health Related Quality of Life | baseline
  Quality of life will be measured using the Minnesota Living with Heart Failure Questionnaire (MLHFQ). Each item is scored in a 6-point Likert Scale (0 to 5), thus the total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life
Health Related Quality of Life | 3-months
  Quality of life will be measured using the Minnesota Living with Heart Failure Questionnaire (MLHFQ). Each item is scored in a 6-point Likert Scale (0 to 5), thus the total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life
Health Related Quality of Life | 6-months
  Quality of life will be measured using the Minnesota Living with Heart Failure Questionnaire (MLHFQ). Each item is scored in a 6-point Likert Scale (0 to 5), thus the total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life
Health Related Quality of Life | 12-months
  Quality of life will be measured using the Minnesota Living with Heart Failure Questionnaire (MLHFQ). Each item is scored in a 6-point Likert Scale (0 to 5), thus the total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life
Health Related Quality of Life | 18-months
  Quality of life will be measured using the Minnesota Living with Heart Failure Questionnaire (MLHFQ). Each item is scored in a 6-point Likert Scale (0 to 5), thus the total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life
Healthcare Utilization | baseline
  Healthcare utilization was determined by the frequency of emergency department visits and readmissions for HF and assessed via self-report.
Healthcare Utilization | 3-months
  Healthcare utilization was determined by the frequency of emergency department visits and readmissions for HF and assessed via self-report.
Healthcare Utilization | 6-months
  Healthcare utilization was determined by the frequency of emergency department visits and readmissions for HF and assessed via self-report.
Healthcare Utilization | 12-months
  Healthcare utilization was determined by the frequency of emergency department visits and readmissions for HF and assessed via self-report.
Healthcare Utilization | 18-months
  Healthcare utilization was determined by the frequency of emergency department visits and readmissions for HF and assessed via self-report.
Stress | baseline
  The Perceived Stress Scale (PSS) will measure perceptions of stress and anger. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived. stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress.
Stress | 3-months
  The Perceived Stress Scale (PSS) will measure perceptions of stress and anger. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived. stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress
Stress | 6-months
  The Perceived Stress Scale (PSS) will measure perceptions of stress and anger. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived. stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress
Stress | 12-months
  The Perceived Stress Scale (PSS) will measure perceptions of stress and anger. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived. stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress
Stress | 18-months
  The Perceived Stress Scale (PSS) will measure perceptions of stress and anger. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived. stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress
Resilience | baseline
  The Five-by-Five Resilience Scale will measure aspects of resilience. Higher scores indicate more resilience.
Resilience | 3-months
  The Five-by-Five Resilience Scale will measure aspects of resilience. Higher scores indicate more resilience.
Resilience | 6-months
  The Five-by-Five Resilience Scale will measure aspects of resilience. Higher scores indicate more resilience.
Resilience | 12-months
  The Five-by-Five Resilience Scale will measure aspects of resilience. Higher scores indicate more resilience.
Resilience | 18-months
  The Five-by-Five Resilience Scale will measure aspects of resilience. Higher scores indicate more resilience.
Coping | baseline
  The Brief COPE will measure the use coping strategies. Each of the 14 scales is comprised of 2 items; total scores on each scale range from 2 (minimum) to 8 (maximum). Higher scores indicate increased utilization of that specific coping strategy. Total scores on each of the scales are calculated by summing the appropriate items for each scale.
Coping | 3-months
  The Brief COPE will measure the use coping strategies. Each of the 14 scales is comprised of 2 items; total scores on each scale range from 2 (minimum) to 8 (maximum). Higher scores indicate increased utilization of that specific coping strategy. Total scores on each of the scales are calculated by summing the appropriate items for each scale.
Coping | 6-months
  The Brief COPE will measure the use coping strategies. Each of the 14 scales is comprised of 2 items; total scores on each scale range from 2 (minimum) to 8 (maximum). Higher scores indicate increased utilization of that specific coping strategy. Total scores on each of the scales are calculated by summing the appropriate items for each scale.
Coping | 12-months
  The Brief COPE will measure the use coping strategies. Each of the 14 scales is comprised of 2 items; total scores on each scale range from 2 (minimum) to 8 (maximum). Higher scores indicate increased utilization of that specific coping strategy. Total scores on each of the scales are calculated by summing the appropriate items for each scale.
Coping | 18-months
  The Brief COPE will measure the use coping strategies. Each of the 14 scales is comprised of 2 items; total scores on each scale range from 2 (minimum) to 8 (maximum). Higher scores indicate increased utilization of that specific coping strategy. Total scores on each of the scales are calculated by summing the appropriate items for each scale.

OTHER OUTCOMES:
Problem-Solving | baseline
  Problem-solving was self-reported and assessed using the Social Problem-Solving Inventory Revised (SPSIR) which measures problem orientation and problem-solving style. In addition to a total score, there are 5 sub-scales: positive problem orientation, negative problem orientation, rational problem-solving, impulsivity/carelessness, and avoidance style. Higher scores on each sub-scale suggest more of the problem-solving characteristic. Higher total scores suggest more adaptive problem-solving, while lower scores indicate more maladaptive problem-solving.
Problem-Solving | 3-months
  Problem-solving was self-reported and assessed using the Social Problem-Solving Inventory Revised (SPSIR) which measures problem orientation and problem-solving style. In addition to a total score, there are 5 sub-scales: positive problem orientation, negative problem orientation, rational problem-solving, impulsivity/carelessness, and avoidance style. Higher scores on each sub-scale suggest more of the problem-solving characteristic. Higher total scores suggest more adaptive problem-solving, while lower scores indicate more maladaptive problem-solving.
Problem-Solving | 6-months
  Problem-solving was self-reported and assessed using the Social Problem-Solving Inventory Revised (SPSIR) which measures problem orientation and problem-solving style. In addition to a total score, there are 5 sub-scales: positive problem orientation, negative problem orientation, rational problem-solving, impulsivity/carelessness, and avoidance style. Higher scores on each sub-scale suggest more of the problem-solving characteristic. Higher total scores suggest more adaptive problem-solving, while lower scores indicate more maladaptive problem-solving.
Problem-Solving | 12-months
  Problem-solving was self-reported and assessed using the Social Problem-Solving Inventory Revised (SPSIR) which measures problem orientation and problem-solving style. In addition to a total score, there are 5 sub-scales: positive problem orientation, negative problem orientation, rational problem-solving, impulsivity/carelessness, and avoidance style. Higher scores on each sub-scale suggest more of the problem-solving characteristic. Higher total scores suggest more adaptive problem-solving, while lower scores indicate more maladaptive problem-solving.
Problem-Solving | 18-months
  Problem-solving was self-reported and assessed using the Social Problem-Solving Inventory Revised (SPSIR) which measures problem orientation and problem-solving style. In addition to a total score, there are 5 sub-scales: positive problem orientation, negative problem orientation, rational problem-solving, impulsivity/carelessness, and avoidance style. Higher scores on each sub-scale suggest more of the problem-solving characteristic. Higher total scores suggest more adaptive problem-solving, while lower scores indicate more maladaptive problem-solving.
Social Support | baseline
  Social support was self-reported and assessed using the Interpersonal Support and Evaluation List - 12 (ISEL-12) which measures perceived belonging, tangible, and appraisal support. Scores range from 0-36, with higher scores suggesting a higher perception of available support.

CONTACTS AND LOCATIONS:
Overall Officials: Lucinda J Graven, PhD, Principal Investigator — Florida State University College of Nursing
Locations (4):
- United States (4):
  - VA Clinic - Gainesville, Gainesville, Florida
  - VA Clinic - Togus, Togus, Maine
  - VA Clinic - Durham, Durham, North Carolina
  - VA Clinic - Providence, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other investigators.

REFERENCES:
- [Derived] Graven LJ, Abbott L, Hodgkins JV, Ledermann T, Howren MB. Supporting Physical and Mental Health in Rural Veterans Living With Heart Failure: Protocol for a Nurse-Led Telephone Intervention Study. JMIR Res Protoc. 2025 Mar 26;14:e63498. doi: 10.2196/63498. PMID 40138689